CLINICAL TRIAL: NCT01490801
Title: Role of the IL-2 Inducible Tcell Kinase in EBV-HLH and EBV+ Hodgkin's Lymphoma
Brief Title: Biomarkers in Blood and Tissue Samples From Patients With Epstein-Barr Virus-Positive Hodgkin Lymphoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AHOD12B1; COG-AHOD12B1 (Other: Children's Oncology Group); AHOD12B1 (Other: Children's Oncology Group); NCI-2012-00089 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Lymphoma; Nonneoplastic Condition
Keywords: childhood Hodgkin lymphoma; childhood mixed cellularity Hodgkin lymphoma; hemophagocytic lymphohistiocytosis; Epstein-Barr virus infection
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphohistiocytosis, Hemophagocytic; Epstein-Barr Virus Infections | interventions — Cytogenetic Analysis; In Situ Hybridization; Polymerase Chain Reaction; Blotting, Western; Flow Cytometry; Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood and Tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: RNA analysis
Genetic: cytogenetic analysis
Genetic: in situ hybridization
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: western blotting
Other: flow cytometry
Other: immunohistochemistry staining method
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies biomarkers in blood and tissue samples from patients with Epstein-Barr virus positive Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate germline DNA from patients with Epstein-Barr virus positive (EBV+) and Hodgkin lymphoma (HL) for inducible T-cell kinase (ITK) mutations.
* Examine the effects of ITK mutations on expression of the ITK protein.
* Determine whether ITK mutations correlate with specific clinical or histopathological features of HL.

OUTLINE: Archived blood and tumor tissue samples are analyzed for germline DNA expression and inducible T-cell kinase (ITK) mutations by PCR, IHC, flow cytometry, and western blotting, and EBV-encoded RNA (EBER) using in situ hybridization. Each patient's data, such as date, sex, age, tumor stage and histology at diagnosis, treatment received, response to treatment, development of recurrent disease, date of last follow-up, and outcomes are also collected.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Hodgkin lymphoma (HL) meeting the following criteria:

  * Epstein-Barr virus-positive (EBV+) HL as assessed by positive EBV serology, elevated levels of EBV genome in the blood or tumor tissue following quantitative polymerase chain reaction (PCR) and/or evidence of EBV positivity of pathology samples (EBER+ or LMP+) and, when possible, mixed cellular histology
  * Young age (< 10 years) at diagnosis
  * Presence of hemophagocytic lymphohistiocytosis (HLH)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Diagnosis of Hodgkin lymphoma.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Presence of germline ITK mutations
Influence of ITK mutations on total expression levels or intracellular localization of the ITK protein
Correlation between ITK mutations with specific clinical or histopathological features of HL

CONTACTS AND LOCATIONS:
Overall Officials: Kim E. Nichols, MD, BA, Principal Investigator — Children's Hospital of Philadelphia